CLINICAL TRIAL: NCT04959682
Title: A Randomized Controlled Pilot Study Evaluating the Effect of Patient-tailored Live Music Interventions for Patients Undergoing Hemodialysis
Brief Title: Music Interventions for Patients Undergoing Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: The Royal Academy of Music Aarhus/Aalborg (Unknown); Aarhus University Hospital (Other); University of Aarhus (Other); Hanze University of Applied Sciences Groningen (Other); University of Music and Performing Arts, Vienna (Unknown); University Hospital of Southern Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Music & Hemodialysis
Record Dates: First submitted 2021-05-26; First posted 2021-07-13 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Renal Failure
Keywords: Music intervention; Feasibility; Kidney failure; Mixed method; Renal dialysis; Randomized Controlled Pilot Study
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will receive 30 minutes of patient-tailored instrumental music in the beginning of one weekly hemodialysis treatment for a period of six weeks
  Interventions: Other: Music Intervention
- Control group (No Intervention): The procedure in the control group is the same as in the intervention group, except that they don't listen to music

INTERVENTIONS:
Other: Music Intervention — After rating levels of fatigue and relaxation, the professional health care musicians will play 30 minutes of patient-tailored, pleasant instrumental music with a combination of relaxing (on average 60-80 bpm) and lively, slightly more up-beat tempo to regulate arousal-levels
  Arms: Intervention group

SUMMARY:
Fatigue is found to be one of the most persistent problems among patients in treatment with hemodialysis, and associated with impaired health-related quality of life. A few, non-randomized controlled trials have found positive effects on fatigue by offering pre-recorded music intra-dialytic, however, without conclusive results. So far, no studies have investigated the feasibility of integrating person-tailored live music interventions performed by professional musicians into a hemodialysis setting. This leaves a deficit in knowledge for intervention planning, understanding and effectiveness of live music on fatigue, wellbeing and feelings of meaningfulness in this group of patients.

Methods: A pilot randomized controlled trial combined with qualitative methods. The data collection will involve recruitment of 24 patients from an outpatient clinic over a six-week period. The patients will be randomized into either an intervention group or a control group. Patients in the intervention group will be offered a 30-minute session of patient-tailored live music intervention per week for six consecutive weeks. Patients in the control group will receive standard care.

Quantitative analysis on immediate post-dialysis fatigue (VAS), and long-term fatigue (MFI-20), anxiety, depression (HADS) and treatment satisfaction (VAS) will show the potential effectiveness of intervention. Qualitative analysis of informal-interviews (patients/staff), observational data (patients) and focus group interviews (staff/musicians) will explore an in-depth understanding of whether music will improve wellbeing and create feelings of meaningfulness among this group of patients as well as to assess feasibility acceptability among patients, musicians and staff.

Perspectives: This trial will ensure a firm methodological approach for the development of a future definitive randomized controlled trial of music intervention for fatigue reduction and wellbeing among hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Scheduled to receive hemodialysis treatment
* Able to understand written and spoken Danish

Exclusion Criteria:

* Deafness
* Severe mental illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Immediate fatigue | Change from baseline immediate fatigue at 8 weeks. VAS is measured at baseline (visit 1), after visit 2, visit 3, visit 4, visit 5, visit 6, visit 7 and at follow-up (visit 8).
  Visual Analogue Scale (VAS). Higher VAS score means higher levels of fatigue
Longterm fatigue | Change from baseline longterm fatigue at 8 weeks. MFI-20 is measured at baseline (visit 1) and at follow-up (visit 8)
  Multidimensional Fatigue Inventory (MFI-20). Higher MFI-20 score means higher levels of fatigue
Post-dialysis fatigue-diary | Change from baseline post dialysis fatigue at 8 weeks. Post-dialysis fatigue is measured the day after visit 2, visit, 3, visit 4, visit 5, visit, 6
  Visual Analogue Scale (VAS). Higher VAS score means higher levels of fatigue

SECONDARY OUTCOMES:
Relaxation | Change from baseline relaxation at 8 weeks. VAS is measured at baseline (visit 1), after visit 2, visit 3, visit 4, visit 5, visit 6, visit 7 and at followup (visit 8)
  Visual Analogue Scale. Higher VAS score means higher levels of relaxation
Anxiety and Depression | Change from baseline anxiety and depression at 8 weeks. HADS is measured at baseline (visit 1) and follow-up (visit 8)
  Hospital Anxiety Depression Scale (HADS). Higher HADS score means higher levels of anxiety and depression
Treatment satisfaction | Change from baseline treatment satisfaction at 8 weeks. VAS is measured at baseline (visit 1) and at follow-up (visit 8)
  Visual Analogue Scale (VAS). Higher VAS score means higher levels of treatment satisfaction
Work engagement (staff) | Change from baseline work engagement at 8 weeks. UWES is measured at baseline (visit 1) and at follow-up (visit 8)
  Utrecht Work Engagement Scale (UWES). Higher UWES score means higher levels of work engagement

CONTACTS AND LOCATIONS:
Overall Officials: Pia Dreyer, PhD, Study Chair — Institute of Public Health, University of Aarhus; Bibi Gram, PhD, Study Chair — Regional Health Research, University of Southern Denmark
Locations (1):
- Margrethe Langer Bro, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No